CLINICAL TRIAL: NCT07162896
Title: Efficacy and Safety of Crisaborole 2% Versus Tacrolimus 0.1% in Children With Mild to Moderate Atopic Dermatitis
Brief Title: Crisaborole 2% Versus Tacrolimus 0.1% in Children With Mild to Moderate Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Kheziema Maryum, Principal Investigator, Shalamar Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kheziema Maryum
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crisaborole 2% Ointment (Active Comparator): Twice daily application to affected areas for 28 days
  Interventions: Drug: Crisaborole 2%
- Tacrolimus 0.1% Ointment (Active Comparator): Twice daily application to affected areas for 28 days
  Interventions: Drug: Tacrolimus 0.1%

INTERVENTIONS:
Drug: Crisaborole 2% — Apply thin layer to affected skin daily for 28 days.
  Arms: Crisaborole 2% Ointment
Drug: Tacrolimus 0.1% — Apply thin layer to affected skin daily for 28 days.
  Arms: Tacrolimus 0.1% Ointment

SUMMARY:
This randomized, open-label, parallel-group study will compare the efficacy and safety of Crisaborole 2% ointment and Tacrolimus 0.1% ointment in children with mild to moderate atopic dermatitis. A total of 66 participants will be randomized (1:1) to receive either Crisaborole or Tacrolimus, applied twice daily to affected areas for 28 days. Primary endpoint is proportion of participants achieving Investigator's Static Global Assessment (ISGA) success (clear/almost clear with ≥2-point improvement from baseline) at Day 28. Safety assessments include adverse events and local application site reactions.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-18 years Both genders Clinically diagnosed mild to moderate atopic dermatitis Body surface area (BSA) <30%

Exclusion Criteria:

Active viral, bacterial, or fungal skin infection at the treatment site

Recent use of topical corticosteroids, calcineurin inhibitors, PDE4 inhibitors, or immunosuppressive medication within past 2 weeks

Known hypersensitivity to study medications or components

Chronic inflammatory conditions (e.g., psoriasis and seborrheic dermatitis) that may interfere with evaluation

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with ISGA sucess ( clear / almost clear from baseline) at day 28. | 28 days
Change in ISGA from baseline to day 28. | Baseline, Day 14, Day 28
  ISGA uses a 5-point scale (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe); negative change indicates improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Shalamar Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No